CLINICAL TRIAL: NCT04052828
Title: Fetal Endoscopic Tracheal Occlusion Trial for Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetal Endoscopic Tracheal Occlusion (FETO) Trial for Congenital Diaphragmatic Hernia (CDH)
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Erin Perrone (Other)
Responsible Party: Sponsor-Investigator, Dr Erin Perrone, Associate Professor of Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00159792
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: pregnant; fetal endoscopic tracheal occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FETO with GOLDBAL2 (Experimental): A balloon will be placed in the airway of the fetus during the FETO procedure.
  Interventions: Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100)

INTERVENTIONS:
Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) — This will take place between gestation of 27w0d - 29w6d. The balloon will be removed at approximately 34 weeks gestation.

SUMMARY:
This is a single site pilot trial to assess the feasibility and safety of treating severe CDH with Fetal Endoscopic Tracheal Occlusion with the Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) at Michigan Medicine. The study will enroll pregnant women that meet study criteria. Participants will have placement of FETO between gestational age at 27 weeks plus 0 days and 29 weeks 6 days. The timing for removal of FETO will ideally be between 34 weeks 0 days and 34 weeks and 6 days but ultimately decided by the Fetal Diagnosis and Treatment Center at Michigan Medicine.

This study requires that study participants live within 30 miles of the Von Voigtlander Women's Hospital and C.S. Mott Children's Hospital in order to maintain weekly follow up appointments while the balloon is in place and up to delivery. Additionally, there are lifestyle considerations where participants would be unable to carry on normal daily activities including exercise and sexual intercourse, not be able to work the remainder of the pregnancy, as well as have a support person that is available to stay with such as a spouse, friend, partner, parent.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Singleton pregnancy
* No pathogenic variants on microarray or pathologic findings on karyotype
* Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects
* Fetal CDH (left or right) with severe pulmonary hypoplasia, defined as observed-to-expected (o/e) lung to head ratios (LHR) <25% with liver up
* Gestational age at FETO procedure: if o/e LHR <25% will be done at 27 weeks plus 0 days to 29 weeks plus 6 days
* Meets psychosocial criteria

  * Willing to reside within 30 minutes of Von Voigtlander Women's Hospital and ability to maintain follow up appointments
  * Patient has a support person (e.g. spouse, partner, friend, parent) that is available to stay with her for the duration of the pregnancy near Von Voigtlander Women's Hospital
  * Willing to comply with restrictions of daily living including inability to exercise, have intercourse, or return to work.

Exclusion Criteria:

* Multi-fetal pregnancy
* History of latex allergy
* History of preterm labor or incompetent cervix (requiring cerclage), short cervix (≤20mm), or uterine anomaly predisposing to preterm labor
* Bilateral CDH, unilateral CDH with o/e LHR > 25%, or unilateral CDH with o/e LHR <25% but liver completely down in abdomen
* Additional fetal or genetic abnormalities that would impact care after delivery or be known to have an impact on outcome
* Maternal contraindications to elective fetoscopic surgery
* Significant placental abnormalities (abruption, chorioangioma, accreta) known at time of enrollment and/or surgery
* Maternal isoimmunization or neonatal alloimmune thrombocytopenia
* Maternal HIV, Hepatitis B with positive surface antigen, Hepatitis C with presence of virus in maternal blood due to risk of fetal transmission during the procedure
* No safe or feasible fetoscopic approach to balloon placement
* Social work will meet with each patient to evaluate the social situation and support system. Identifiable issues of social instability or compliance with the protocol will exclude her as a potential candidate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 10 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of successful placements of the Goldballoon Detachable Balloon (GOLDBAL2) at gestational age 27 weeks zero days (27w0d) to 29 weeks and 6 days (29w6d) gestation. | 27w0d - 29w6d
  Success will be defined as completion with direct visual placement above the carina and confirmation on ultrasound done during the procedure.
Number of successful retrievals of the GOLDBAL2 | Removal prior to delivery approximately 34 weeks of gestation
  This will ideally occur around the 34th week of gestation and have the balloon removed prior to delivery.

SECONDARY OUTCOMES:
Change in observed to expected total fetal lung to head ratios (o/e TFLV) on prenatal magnetic resonance imaging (MRI) | baseline (prior to balloon placement), approximately 2 weeks after balloon retrieval
  Fetal MRI done prior to balloon placement and again done at approximately 2 weeks of balloon retrieval.
Change in fetal lung growth | baseline (before balloon placement), immediately prior to balloon retrieval
  Fetal ultrasounds will be done weekly while the balloon is in place. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR immediately prior to balloon removal.
Gestational age at delivery | At the time of delivery (up to approximately 34 weeks)
Survival of infant to hospital discharge or 180 days after hospitalized | Discharge from hospital or up to 180 days in the hospital
  This will be measured after the infant is delivered to hospital discharge or analyzed for survival at 180 days for those still hospitalized at that time point.
Number of maternal complications | up to 4-6 weeks postpartum
  Complications during pregnancy, and/or at delivery and follow-up to include; preterm labor, premature rupture of membranes (PROM), Preterm Premature Rupture of Membranes (PPROM), oligohydramnios, polyhydramnios, placental abruption, chorioamniotic separation, chorioamnionitis, and other infection.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Perrone, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No